CLINICAL TRIAL: NCT01121263
Title: Hybrid Revascularization Observational Study
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: International Center for Health Outcomes and Innovation Research (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: GCO 09-0657; 1RC1HL100951 (NIH)
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Artery Disease
Keywords: coronary arteriosclerosis; coronary heart disease; coronary artery bypass; coronary artery bypass, off-pump; coronary angiography; drug-eluting stents
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Angiogram Review Group: All consecutive and consenting patients undergoing diagnostic cardiac catheterization in a 3 month period
- Therapeutic Intervention Group: * Cohort 2 Therapeutic Intervention Group - HCR Patients (including those from the angiogram review group) who undergo Hybrid coronary revascularization (HCR) with minimally invasive LIMA-LAD CABG, OR
  * Cohort 2 Therapeutic Intervention Group - PCI Patients (including those from the angiogram review group) who meet the proposed anatomic and clinical eligibility criteria and undergo multivessel Percutaneous Coronary Intervention with Drug Eluting Stents

SUMMARY:
The purpose of the study is to get a better understanding of patients who have multi-vessel coronary artery disease (blockages in more than one vessel bringing blood to the heart) and have either Hybrid Coronary Revascularization [HCR] (combination of surgery and catheter procedures to open up clogged heart arteries) or Percutaneous Coronary Intervention [PCI] (catheter procedures to open up clogged heart arteries). Participation in the study will last up to 21 months after a patient's heart procedure(s). The study collects information about the medical care patients receive during their planned procedure(s) and how well they do following the procedure(s). No new testing or procedures will be done. Patients will receive only the tests or procedures their doctor already has planned for them. The information collected should help to plan the design of a pivotal comparative effectiveness study of hybrid revascularization.

DETAILED DESCRIPTION:
The increasing prevalence of coronary artery disease (CAD), advances in coronary artery bypass grafting (CABG), percutaneous coronary intervention (PCI), and concomitant medical therapy, and the costs of revascularization have resulted in rising interest regarding the appropriate indications for coronary revascularization. For patients with 3-vessel disease, revascularization by CABG has recently been rated as appropriate while revascularization by PCI has been rated uncertain. Ideally, physicians would like to offer their multi-vessel CAD patients what they truly seek: a solution which provides a safe, minimally invasive treatment that does not compromise long term durability and survival. Integrating the positive features of both PCI and CABG has been the fundamental rationale of "hybrid" coronary revascularization.

Hybrid Coronary Revascularization (HCR) (the intended combination of CABG and PCI) as a scientifically validated approach would have a major healthcare impact. The ability to deliver a new therapy for CAD that provides durability, but without the obligatory trauma and prolonged recovery time characteristic of conventional CABG would be a major advance in the field of cardiovascular medicine. Candidates in whom HCR would be particularly advantageous would be several subgroups of CAD patients that are increasing in numbers: the elderly, patients with a high predicted risk of mortality and/or morbidity for CABG, deconditioned patients or patients with significant disabilities and patients in whom treatment durability is important, but a significantly invasive approach is not an option. Moreover, HCR is likely to bridge the divide in treatment philosophies and approaches that exist between cardiologists and cardiac surgeons. Collaboration rather than competition between these specialties will ultimately benefit patients, hospitals, payers and healthcare providers. The Hybrid Revascularization Observational Study is a multi-center observational study planning grant which will explore target populations for Hybrid Coronary Revascularization (HCR), their outcomes, and variations in specific ways these patients are managed, in order to inform the design of a pivotal comparative effectiveness trial of this emerging therapeutic strategy.

Given the observational nature of the study, the HCR and PCI groups' baseline characteristics and event rates are not directly comparable; rather, the results were intended to inform the design of a larger, randomized pivotal trial. The study was designed in two phases: Cohort 1, which captured demographic, angiographic, and practice patterns data for 6,669 consecutively screened patients; and Cohort 2 which captured demographic, angiographic, practice patterns, and outcome data for 298 patients who underwent either HCR or PCI with DES (90 of whom were also part of Cohort 1).

ELIGIBILITY:
The following criteria apply to Cohort 2 PCI patients only:

Inclusion Criteria:

* Signed informed consent, release of medical information, and Health Insurance Portability and Accountability Act (HIPAA) documents
* Age 18 years or older
* Clinical indication for revascularization
* LAD and at least one additional vessel coronary disease (> 70% stenosis) confirmed by angiogram
* Clinical characteristics and multi-vessel disease amenable to both PCI with DES and Hybrid as adjudicated by one interventional cardiologist and one cardiac surgeon
* Ability to tolerate and no plans to interrupt double platelet therapy for ≥ 12 months
* Ability to tolerate to single lung ventilation in the judgment of the investigator
* Willing to comply with all protocol required follow-up

Exclusion Criteria:

* Previous coronary stent within:

  * 1 month prior to enrollment for bare metal stent (BMS) or
  * 6 months prior to enrollment for DES
* Evidence of in stent restenosis of a DES or BMS
* Previous cardiac surgery of any kind
* Chronic total occlusion (CTO) in LAD or ≥ 2 CTOs in major coronary territories that are considered targets for revascularization
* Left main disease ≥ 50% stenosis
* Presence of fresh coronary thrombus
* Need for concomitant vascular or other cardiac surgery during the index hospitalization (including, but not limited to, valve surgery, aortic resection, left ventricular aneurysm, carotid endarterectomy or stenting, etc)
* Previous STEMI within 30 days prior to randomization
* Previous stroke within 6 months prior to randomization
* Previous thoracic surgery involving the left pleural space
* Acute decompensated heart failure within 30 days prior to randomization
* Ejection fraction < 30%
* Creatinine clearance ≤ 50 ml/min within 24 hours prior to randomization
* Hemodynamic instability at time of screening
* Body mass index > 40
* Extra-cardiac illness that is expected to limit survival to less than 3 years
* Participation or planned participation in another investigational intervention study within 60 days prior to randomization
* Unable to give informed consent or potential for noncompliance with the study protocol due to psychiatric illness, organic brain disease, dementia, current alcohol abuse, mental retardation, language barrier, or geographical inaccessibility;
* Pregnancy at time of screening or intention to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1 (Angiogram Review Group): All consecutive and consenting patients undergoing diagnostic cardiac catheterization in a 3 month period.
  Cohort 2 (Therapeutic Intervention Group): All patients (including those from cohort 1) who meet either of the following: (a) undergo HCR with minimally invasive LIMA-LAD CABG (HCR Group) OR (b) meet the proposed anatomic and clinical eligibility criteria defined below and undergo multivessel PCI with DES (PCI Group).
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Puskas, MD, MSc, FACS, FACC, Principal Investigator — Emory University; Deborah Ascheim, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai (Data Coordinating Center); Joseph J DeRose, MD, FACS, Principal Investigator — Montefiore Medical Center; Michael Argenziano, MD, FACS, Principal Investigator — Columbia University; Mathew Williams, MD, Principal Investigator — Columbia University; John G. Byrne, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (11):
- United States (11):
  - Emory University, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Virginia Health Systems, Charlottesville, Virginia

REFERENCES:
- [Derived] Puskas JD, Halkos ME, DeRose JJ, Bagiella E, Miller MA, Overbey J, Bonatti J, Srinivas VS, Vesely M, Sutter F, Lynch J, Kirkwood K, Shapiro TA, Boudoulas KD, Crestanello J, Gehrig T, Smith P, Ragosta M, Hoff SJ, Zhao D, Gelijns AC, Szeto WY, Weisz G, Argenziano M, Vassiliades T, Liberman H, Matthai W, Ascheim DD. Hybrid Coronary Revascularization for the Treatment of Multivessel Coronary Artery Disease: A Multicenter Observational Study. J Am Coll Cardiol. 2016 Jul 26;68(4):356-65. doi: 10.1016/j.jacc.2016.05.032. PMID 27443431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Recruitment started in May 2010 and completed in November 2011 across 11 US medical centers that included adult patients with multivessel coronary artery disease and clinical indication for revascularization, who were candidates for both Hybrid Coronary Revascularization (HCR) and Percutaneous Coronary Intervention (PCI) with DES
Groups:
- Cohort 2: Intervention Cohort - HCR Group (N=200): Patients who underwent Hybrid Coronary Revascularization (HCR) with minimally invasive LIMA-LAD CABG
- Cohort 2: Intervention Cohort - PCI Group (N=98): Patients who met proposed anatomic and clinical eligibility criteria and underwent multivessel Percutaneous Coronary Intervention (PCI) with drug eluting stents (DES)
Period: Overall Study
Arm/Group | Cohort 2: Intervention Cohort - HCR Group (N=200) | Cohort 2: Intervention Cohort - PCI Group (N=98)
Started | 200 | 98
Completed | 175 | 83
Not Completed | 25 | 15
Not completed — Death | 3 | 2
Not completed — Lost to Follow-up | 22 | 12
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 2: Intervention Cohort - HCR Group (N=200) | Cohort 2: Intervention Cohort - PCI Group (N=98) | Total
Number analyzed (Participants) | 200 | 98 | 298
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 64.41 (11.78) | 63.91 (10.82) | 64.24 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 28 | 76
  Male | 152 | 70 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 183 | 83 | 266
  Unknown or Not Reported | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 28 | 11 | 39
  White | 161 | 83 | 244
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 200 | 98 | 298

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiac and Cerebrovascular Event (MACCE)
Description: For the purposes of this study MACCE is defined as a non-weighted composite score comprised of the following components:
  * Death
  * Stroke
  * Myocardial Infarction
  * Repeat Revascularization
Time Frame: Month 12
Measure: Number; unit: participants
Groups:
- HCR Group (N=200): Primary Outcome in Cohort 2: Intervention Cohort - HCR Group
- PCI Group (N=98): Primary Outcome in Cohort 2: Intervention Cohort - PCI Group
Arm/Group | HCR Group (N=200) | PCI Group (N=98)
Number analyzed (Participants) | 200 | 98
participants
  Any MACCE | 23 [0.666 to 1.697] | 10
  Death | 3 [0.666 to 1.697] | 1
  Myocardial Infarction | 4 [0.666 to 1.697] | 3
  Stroke | 5 [0.666 to 1.697] | 0
  Revascularization | 14 [0.666 to 1.697] | 8
Statistical Analysis 1: Comparison: HCR Group (N=200) vs PCI Group (N=98); This applies to any MACCE; Test type: Superiority or Other; p = 0.80, Regression, Cox; The Cox proportional hazards regression model was weighted by propensity score to adjust for differences in baseline risk between the two groups; Hazard Ratio (HR) = 1.063, 95% CI [0.666 to 1.697] — The Cox model was weighted by propensity score to adjust for differences in baseline risk between the two groups

2. Secondary Outcome: Major Adverse Cardiac and Cerebrovascular Event (MACCE)
Description: as for outcome 1
Time Frame: Occurence of MACCE through the end of study up to two years
Measure: Number; unit: participants
Groups:
- HCR Group (N=200): Occurrence of MACCE through the end of study in Cohort 2: Intervention Cohort - HCR Group
- PCI Group (N=98): Occurrence of MACCE through the end of study in Cohort 2: Intervention Cohort - PCI Group
Arm/Group | HCR Group (N=200) | PCI Group (N=98)
Number analyzed (Participants) | 200 | 98
participants
  Any MACCE | 23 | 12
  Death | 3 | 2
  Myocardial Infarction | 4 | 3
  Stroke | 5 | 0
  Revascularization | 14 | 10
Statistical Analysis 1: Comparison: HCR Group (N=200) vs PCI Group (N=98); This applies to any MACCE; Test type: Superiority or Other; p = 0.53, Regression, Cox; Hazard Ratio (HR) = 0.868, 95% CI [0.556 to 1.355] — The Cox proportional hazards regression model was weighted by the propensity score to account for the difference in baseline risk between groups

ADVERSE EVENTS:
Time Frame: Adverse events were reported throughout the period of trial participation for each study participant.
Description: Adverse events were documented and reported by staff at the study sites as they occurred per the protocol definitions.
Groups:
- HCR Group (N=200): Serious Adverse Events in Cohort 2: Intervention Cohort - HCR Group
- PCI Group (N=98): Serious Adverse Events in Cohort 2: Intervention Cohort - PCI Group
Arm/Group | HCR Group (N=200) | PCI Group (N=98)
Serious Adverse Events (participants affected / at risk) | 39/200 | 17/98
Other Adverse Events (participants affected / at risk) | 5/200 | 0/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCR Group (N=200) (N=200) | PCI Group (N=98) (N=98)
Cardiac Arrhythmias (Cardiac disorders) | 6 (6) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (2) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1)
Diastolic Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Dresseler's Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension Resulting in Dizziness (Cardiac disorders) | 1 (1) | 0 (0)
IABP placed after becoming hypotensive (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 3 (4) | 3 (4)
Revascularization (Cardiac disorders) | 13 (14) | 10 (12)
Acute viral gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI Bleed (Gastrointestinal disorders) | 2 (2) | 0 (0)
Allergic reaction to antihypertensive drug (General disorders) | 1 (1) | 0 (0)
Atypical Chest Pain (General disorders) | 1 (1) | 5 (5)
Bleeding (General disorders) | 1 (1) | 0 (0)
Weakness and dizziness (General disorders) | 0 (0) | 1 (1)
Major Infection (Infections and infestations) | 6 (6) | 0 (0)
Stroke (Nervous system disorders) | 4 (4) | 0 (0)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 2 (2) | 0 (0)
Post op deliriums/psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia with bladder obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Percutaneous transluminal angioplasty of superficial femoral artery (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCR Group (N=200) (N=200) | PCI Group (N=98) (N=98)
Cardiac Arrhythmias (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Revascularization (Cardiac disorders) | 1 (1) | 0 (0)
Major Infection (Infections and infestations) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MSSM and sites shall cooperate in the submission of manuscript(s) for publication of the study results and sites shall not submit manuscripts for publication without express written permission of the Operations Committee. After dissolution of the Operations committee or one year after the completion of the agreement, whichever occurs first, no such permission shall be required.